CLINICAL TRIAL: NCT06718400
Title: Vascularised Sentinel Skin Flaps to Predict Rejection in Intestinal Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of PI
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anil Vaidya, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-882
Record Dates: First submitted 2022-05-09; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Intestinal Transplant
Keywords: Transplant; Sentinel Skin Flap

STUDY DESIGN:
Intervention Model Description: Willing participants who will be receiving an intestinal transplantation will receive a sentinel skin flap on their forearm from the same donor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Skin Flap (Experimental): Willing participants who will be receiving an intestinal transplantation will receive a sentinel skin flap on their forearm from the same donor
  Interventions: Procedure: Sentinel Skin Flap

INTERVENTIONS:
Procedure: Sentinel Skin Flap — Willing participants who will be receiving an intestinal transplantation will receive a sentinel skin flap on their forearm from the same donor

SUMMARY:
This pilot study aims to validate the use of vascularised donor-derived sentinel skin flaps for diagnosing and monitoring rejection in intestinal transplantation

DETAILED DESCRIPTION:
Intestinal transplantation is the current treatment option for patients with irreversible intestinal failure that has not responded to other methods of treatment. Whilst the majority of patients that have an intestinal transplant will obtain good graft function over many years, some patients suffer from reduced function of their new intestine following transplantation that can progress to the transplant failing completely.

Acute rejection may be the most common cause of transplant failure. Currently, there is not an effective way of monitoring the intestine that can detect rejection before irreversible damage occurs. If there is a more sensitive way of continuously monitoring the intestine transplant for rejection then issues could be earlier detected and early treatment could prevent permanent damage to the transplant.

The reason for this study is to assess a new technique that has been developed to detect early rejection in intestinal transplantation. The name of this technique is called a 'sentinel skin flap' and involves transplanting a patch of forearm skin from the donor at the same time as the intestine

ELIGIBILITY:
Inclusion Criteria

* Recipient of an intestinal transplant.
* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above

Exclusion Criteria

* Patient does not have a patent ulnar artery in either forearm or a negative Allen's test.
* Patient is not willing to return to the Institution for all clinical follow-up for 12 months
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the trial, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of histological rejection in the skin flap and the transplanted solid organ | 12 months
  To establish if a sentinel skin flap acts as a marker of rejection of the transplanted organ.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Vaidya, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No